CLINICAL TRIAL: NCT01986439
Title: The Contraceptive Choice Project
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jeffrey Peipert, Robert J. Terry Professor, Washington University School of Medicine
Other Study IDs: 201101982
Record Dates: First submitted 2013-10-31; First posted 2013-11-18 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Unintended Pregnancy; Teen Births; Abortion; Contraception

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — vaginal swab specimens for chlamydia, gonorrhea, trichomoniasis, and bacterial vaginosis. Blood specimens for HIV and syphilis.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this project is to remove barriers to obtaining contraceptive methods, including the most effective and expensive methods. The study seeks to remove the financial and knowledge barriers and promote the most effective contraceptive methods to reduce unintended pregnancy rates at the population level.

ELIGIBILITY:
Inclusion Criteria:

1. 14-45 years of age
2. Primary residency in St. Louis City or County
3. Does not desire pregnancy during the next 1 year
4. Desires reversible contraception
5. Sexually active with a man within the past 6 months or intend to have sex with a man in the next 6 months
6. Is not currently using a contraceptive method, has begun using a new contraceptive method within the last 4 weeks, or is a current contraceptive method user who wants to switch to a NEW contraceptive method immediately
7. Willing and able to undergo informed consent
8. Willing to comply with study protocol and 2-year follow-up schedule
9. Not currently pregnant, or meets one of the following criteria:

   1. Currently pregnant, undergoing medical or surgical termination of pregnancy, and planning for post-abortion contraception
   2. Currently pregnant with an abnormal pregnancy (miscarriage or ectopic pregnancy), undergoing medical or surgical management, and planning for post-pregnancy contraception
   3. Currently pregnant, estimated gestational age of 36 weeks or greater, and planning for post-partum contraception.

Exclusion Criteria:

1. History of hysterectomy or sterilization
2. Current participation in another research study that would interfere with the conduct of this study

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women of reproductive age who reside in the St. Louis metropolitan region.
Sampling Method: Non-Probability Sample
Enrollment: 9256 (Actual)
Dates: Start 2007-08; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Distribution of contraceptive method chosen | Baseline
  Distribution of methods (%) chosen at baseline enrollment, by method and stratified by Long-Acting Reversible Contraception (LARC: intrauterine device and implant) and non-LARC (depotmedroxyprogesterone acetate (DMPA), oral contraceptive pill (OCP), vaginal ring, transdermal patch).

SECONDARY OUTCOMES:
Method Continuation | 6-month, 12 month, 24-month, and 36-month
  % of women using each method at 6, 12-, 24, and 36 months post-enrollment. Hazard rates via survival analysis comparing LARC and non-LARC methods.
Method Satisfaction | 12-month, 24-month, 36-month
  % of women very or somewhat satisfied with method at 12, 24, and 36 months of use. Comparison of all methods and stratified by LARC and non-LARC methods.
Teen Pregnancy Rates | 1-year, 2-year, 3-year
  Number of pregnancies per participants 15-19 years of age. We will calculate an annual rate for each year from 2007-2013 and also calculate a rate for the cohort followed for 1 year, 2 years, and 3 years.
Repeat Abortion Rates | 1-year, 2-year, 3-year
  Number of abortions among participants 15-44 with a history of abortion. We will calculate an annual rate for each year from 2007-2013 and also calculate a rate for the cohort followed for 1 year, 2 years, and 3 years.
Sexually transmitted infection rates | Baseline and 12-months
  Baseline prevalence rates (number positive divided by number tested) for chlamydia, gonorrhea, and trichomonas. 1-year incidence rates for the same infections among those who tested at 1-year.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey F Peipert, MD PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Result] Tepe M, Mestad R, Secura G, Allsworth JE, Madden T, Peipert JF. Association between tampon use and choosing the contraceptive vaginal ring. Obstet Gynecol. 2010 Apr;115(4):735-739. doi: 10.1097/AOG.0b013e3181d41c4a. PMID 20308832
- [Result] Secura GM, Allsworth JE, Madden T, Mullersman JL, Peipert JF. The Contraceptive CHOICE Project: reducing barriers to long-acting reversible contraception. Am J Obstet Gynecol. 2010 Aug;203(2):115.e1-7. doi: 10.1016/j.ajog.2010.04.017. Epub 2010 Jun 11. PMID 20541171
- [Result] Spain JE, Peipert JF, Madden T, Allsworth JE, Secura GM. The Contraceptive CHOICE Project: recruiting women at highest risk for unintended pregnancy and sexually transmitted infection. J Womens Health (Larchmt). 2010 Dec;19(12):2233-8. doi: 10.1089/jwh.2010.2146. Epub 2010 Sep 11. PMID 20831439
- [Result] Pittman ME, Secura GM, Allsworth JE, Homco JB, Madden T, Peipert JF. Understanding prescription adherence: pharmacy claims data from the Contraceptive CHOICE Project. Contraception. 2011 Apr;83(4):340-5. doi: 10.1016/j.contraception.2010.08.003. Epub 2010 Sep 17. PMID 21397092
- [Result] Peipert JF, Zhao Q, Allsworth JE, Petrosky E, Madden T, Eisenberg D, Secura G. Continuation and satisfaction of reversible contraception. Obstet Gynecol. 2011 May;117(5):1105-1113. doi: 10.1097/AOG.0b013e31821188ad. PMID 21508749
- [Result] Kittur ND, Secura GM, Peipert JF, Madden T, Finer LB, Allsworth JE. Comparison of contraceptive use between the Contraceptive CHOICE Project and state and national data. Contraception. 2011 May;83(5):479-85. doi: 10.1016/j.contraception.2010.10.001. Epub 2010 Nov 23. PMID 21477693
- [Result] Kossler K, Kuroki LM, Allsworth JE, Secura GM, Roehl KA, Peipert JF. Perceived racial, socioeconomic and gender discrimination and its impact on contraceptive choice. Contraception. 2011 Sep;84(3):273-9. doi: 10.1016/j.contraception.2011.01.004. Epub 2011 Feb 21. PMID 21843693
- [Result] Mestad R, Secura G, Allsworth JE, Madden T, Zhao Q, Peipert JF. Acceptance of long-acting reversible contraceptive methods by adolescent participants in the Contraceptive CHOICE Project. Contraception. 2011 Nov;84(5):493-8. doi: 10.1016/j.contraception.2011.03.001. Epub 2011 Apr 27. PMID 22018123
- [Result] Graseck AS, Secura GM, Allsworth JE, Madden T, Peipert JF. Home screening compared with clinic-based screening for sexually transmitted infections. Obstet Gynecol. 2010 Apr;115(4):745-752. doi: 10.1097/AOG.0b013e3181d4450d. PMID 20308834
- [Result] Graseck AS, Secura GM, Allsworth JE, Madden T, Peipert JF. Home compared with clinic-based screening for sexually transmitted infections: a randomized controlled trial. Obstet Gynecol. 2010 Dec;116(6):1311-1318. doi: 10.1097/AOG.0b013e3181fae60d. PMID 21099596
- [Result] Shih SL, Kebodeaux CA, Secura GM, Allsworth JE, Madden T, Peipert JF. Baseline correlates of inconsistent and incorrect condom use among sexually active women in the contraceptive CHOICE Project. Sex Transm Dis. 2011 Nov;38(11):1012-9. doi: 10.1097/OLQ.0b013e318225f8c3. PMID 21992976
- [Result] Madden T, Secura GM, Allsworth JE, Peipert JF. Comparison of contraceptive method chosen by women with and without a recent history of induced abortion. Contraception. 2011 Dec;84(6):571-7. doi: 10.1016/j.contraception.2011.03.018. Epub 2011 May 4. PMID 22078185
- [Result] Madden T, Proehl S, Allsworth JE, Secura GM, Peipert JF. Naproxen or estradiol for bleeding and spotting with the levonorgestrel intrauterine system: a randomized controlled trial. Am J Obstet Gynecol. 2012 Feb;206(2):129.e1-8. doi: 10.1016/j.ajog.2011.09.021. Epub 2011 Sep 24. PMID 22055339
- [Result] Madden T, Grentzer JM, Secura GM, Allsworth JE, Peipert JF. Risk of bacterial vaginosis in users of the intrauterine device: a longitudinal study. Sex Transm Dis. 2012 Mar;39(3):217-22. doi: 10.1097/OLQ.0b013e31823e68fe. PMID 22337109
- [Result] Skala SL, Secura GM, Peipert JF. Factors associated with screening for sexually transmitted infections. Am J Obstet Gynecol. 2012 Apr;206(4):324.e1-6. doi: 10.1016/j.ajog.2012.02.020. Epub 2012 Feb 28. PMID 22464074
- [Result] Winner B, Peipert JF, Zhao Q, Buckel C, Madden T, Allsworth JE, Secura GM. Effectiveness of long-acting reversible contraception. N Engl J Med. 2012 May 24;366(21):1998-2007. doi: 10.1056/NEJMoa1110855. PMID 22621627
- [Result] Peipert JF, Madden T, Allsworth JE, Secura GM. Preventing unintended pregnancies by providing no-cost contraception. Obstet Gynecol. 2012 Dec;120(6):1291-7. doi: 10.1097/aog.0b013e318273eb56. PMID 23168752
- [Result] Secura GM, Desir FA, Mullersman JL, Madden T, Allsworth JE, Peipert JF. Predictors of male partner treatment for sexually transmitted infection. Sex Transm Dis. 2012 Oct;39(10):769-75. doi: 10.1097/OLQ.0b013e31825ec611. PMID 23001263
- [Result] McNicholas C, Peipert JF, Maddipati R, Madden T, Allsworth JE, Secura GM. Sexually transmitted infection prevalence in a population seeking no-cost contraception. Sex Transm Dis. 2013 Jul;40(7):546-51. doi: 10.1097/OLQ.0b013e31829529eb. PMID 23965768
- [Result] Eisenberg DL, Secura GM, Madden TE, Allsworth JE, Zhao Q, Peipert JF. Knowledge of contraceptive effectiveness. Am J Obstet Gynecol. 2012 Jun;206(6):479.e1-9. doi: 10.1016/j.ajog.2012.04.012. Epub 2012 Apr 6. PMID 22521458
- [Result] Madden T, Mullersman JL, Omvig KJ, Secura GM, Peipert JF. Structured contraceptive counseling provided by the Contraceptive CHOICE Project. Contraception. 2013 Aug;88(2):243-9. doi: 10.1016/j.contraception.2012.07.015. Epub 2012 Sep 5. PMID 22959396
- [Result] Xu H, Wade JA, Peipert JF, Zhao Q, Madden T, Secura GM. Contraceptive failure rates of etonogestrel subdermal implants in overweight and obese women. Obstet Gynecol. 2012 Jul;120(1):21-6. doi: 10.1097/AOG.0b013e318259565a. PMID 22678035
- [Result] Rosenstock JR, Peipert JF, Madden T, Zhao Q, Secura GM. Continuation of reversible contraception in teenagers and young women. Obstet Gynecol. 2012 Dec;120(6):1298-305. doi: 10.1097/aog.0b013e31827499bd. PMID 23168753
- [Result] Nault AM, Peipert JF, Zhao Q, Madden T, Secura GM. Validity of perceived weight gain in women using long-acting reversible contraception and depot medroxyprogesterone acetate. Am J Obstet Gynecol. 2013 Jan;208(1):48.e1-8. doi: 10.1016/j.ajog.2012.10.876. Epub 2012 Oct 24. PMID 23103344
- [Result] Stuart JE, Secura GM, Zhao Q, Pittman ME, Peipert JF. Factors associated with 12-month discontinuation among contraceptive pill, patch, and ring users. Obstet Gynecol. 2013 Feb;121(2 Pt 1):330-336. doi: 10.1097/AOG.0b013e31827e5898. PMID 23344283
- [Result] Vickery Z, Madden T, Zhao Q, Secura GM, Allsworth JE, Peipert JF. Weight change at 12 months in users of three progestin-only contraceptive methods. Contraception. 2013 Oct;88(4):503-8. doi: 10.1016/j.contraception.2013.03.004. Epub 2013 Mar 18. PMID 23582238
- [Result] O'Neil-Callahan M, Peipert JF, Zhao Q, Madden T, Secura G. Twenty-four-month continuation of reversible contraception. Obstet Gynecol. 2013 Nov;122(5):1083-1091. doi: 10.1097/AOG.0b013e3182a91f45. PMID 24104781
- [Result] Grunloh DS, Casner T, Secura GM, Peipert JF, Madden T. Characteristics associated with discontinuation of long-acting reversible contraception within the first 6 months of use. Obstet Gynecol. 2013 Dec;122(6):1214-21. doi: 10.1097/01.AOG.0000435452.86108.59. PMID 24201685
- [Result] McNicholas CP, Madden T, Zhao Q, Secura G, Allsworth JE, Peipert JF. Cervical lidocaine for IUD insertional pain: a randomized controlled trial. Am J Obstet Gynecol. 2012 Nov;207(5):384.e1-6. doi: 10.1016/j.ajog.2012.09.018. Epub 2012 Sep 20. PMID 23107081
- [Derived] Leroy-Melamed M, Zhao Q, Belmonte MA, Archer J, Peipert JF. Contraceptive Preference, Continuation Rates, and Unintended Pregnancies in Patients with Comorbidities: A Prospective Cohort Study. J Womens Health (Larchmt). 2021 Oct;30(10):1469-1475. doi: 10.1089/jwh.2020.8536. Epub 2021 Jan 6. PMID 33404367
- [Derived] Bernard C, Zhao Q, Peipert JF. Dual method use among long-acting reversible contraceptive users. Eur J Contracept Reprod Health Care. 2018 Apr;23(2):97-104. doi: 10.1080/13625187.2018.1445850. Epub 2018 Mar 27. PMID 29582687
- See also: CHOICE Project Website — http://www.choiceproject.wustl.edu